CLINICAL TRIAL: NCT02821923
Title: Effect of the Natural Sweeteners Erythritol and Xylitol on Vascular Function in Obese Volunteers: A Pilot Study
Brief Title: Effect of the Natural Sweeteners Erythritol and Xylitol on Vascular Function in Obese Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Poly Vasc
Record Dates: First submitted 2016-06-27; First posted 2016-07-04 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): no treatment
- E967-Xylitol (Active Comparator): 24g xylitol/d
  Interventions: Dietary Supplement: E967-Xylitol
- E968-Erythritol (Active Comparator): 36g erythritol/d
  Interventions: Dietary Supplement: E968-Erythritol

INTERVENTIONS:
Dietary Supplement: E967-Xylitol — 24g xylitol/d
  Arms: E967-Xylitol
Dietary Supplement: E968-Erythritol — 36g erythritol/d
  Arms: E968-Erythritol

SUMMARY:
Sugar alcohols such as xylitol and erythritol are increasingly popular as sugar substitutes in the food industry and are also recommended to diabetic patients. Both substances are already in use in the food industry and are freely available. Since the 1970s, beneficial effects on oral health could be demonstrated as oral bacteria were influenced positively. A pilot study recently undertaken in the US (Flint N, 2014) has shown that diabetics profit from a daily intake of erythritol, as this natural sweetener enhances the elasticity of the blood vessels. In this trial, investigators aim to examine whether this effect can be found in a non-diabetic but obese cohort, and whether also xylitol improves vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Obese volunteers (BMI > 30kg/m2)
* Aged 18- max. 55 years
* Otherwise healthy.

Exclusion Criteria:

* Known cardiovascular disease
* Diabetes mellitus
* Smoking and drug abuse
* Arterial hypertension with antihypertensive treatment
* Dyslipidaemia with statin therapy
* Known chronic hepatic disease (NASH, hepatitis).
* Known renal disease: kidney failure
* Pregnancy
* Chronical diseases of the gastrointestinal tract, history of gastrointestinal surgery with major changes to the gastrointestinal tract
* Substance abuse, alcohol abuse.
* Inability to follow procedures due to psychological disorders, dementia or insufficient knowledge of project language (German).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Central arterial stiffness measured by sonography | Change from baseline to 5 weeks after intake of polyol

SECONDARY OUTCOMES:
Glucose tolerance measured by oral glucose tolerance test | Change from baseline to 5 weeks after intake of polyol

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Study Chair — St. Claraspital Basel klinische Forschungsabteilung
Locations (1):
- University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bordier V, Teysseire F, Drewe J, Madorin P, Bieri O, Schmidt-Trucksass A, Hanssen H, Beglinger C, Meyer-Gerspach AC, Wolnerhanssen BK. Effects of a 5-week intake of erythritol and xylitol on vascular function, abdominal fat and glucose tolerance in humans with obesity: a pilot trial. BMJ Nutr Prev Health. 2023 Nov 14;6(2):264-272. doi: 10.1136/bmjnph-2023-000764. eCollection 2023. PMID 38618550